CLINICAL TRIAL: NCT01580163
Title: Efficacy Evaluation of Traditional Chinese Medicine JITAI Combined Comprehensive Model Among Heroin Addicts After Detoxification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Center of Biomedicine Development (Unknown)
Responsible Party: Principal Investigator, Min ZHAO, vise president, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MZhao-002
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Heroin Addiction
Keywords: the opioid dependence in rehabilitation phase; community
MeSH Terms: conditions — Heroin Dependence | interventions — Psychosocial Intervention; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- JITAI combined therapy group (Experimental): The investigator will adopt JITAI combined psychological intervention and social support in Shanghai-related community.
  Interventions: Drug: JITAI Combined with psychological intervention
- Methadone combined herapy group (Experimental): The investigator will adopt JITAI combined psychological intervention and social support in Shanghai-related community.
  Interventions: Drug: Methadone
- JITAI therapy group (Experimental): The investigator will adopt JITAI combined social support in Shanghai-related community and outside of Shanghai.
  Interventions: Drug: Traditional Chinese Medicine JITAI

INTERVENTIONS:
Drug: JITAI Combined with psychological intervention — tablet，Each tablet weight 0.4g
  Arms: JITAI combined therapy group
Drug: Methadone — Oral Solution，1mg/ml
  Arms: Methadone combined herapy group
Drug: Traditional Chinese Medicine JITAI — tablet，Each tablet weight 0.4g
  Other Names: JITAI
  Arms: JITAI therapy group

SUMMARY:
The purpose of this research is to observe the efficacy of comprehensive treatment model to improve treatment compliance and relapse prevention.

DETAILED DESCRIPTION:
The model include the Chinese traditional medicine JITAI combined with psychological intervention and social support for maintenance therapy after acute detoxification of heroin addicts.On the basis of the existing community management experience and community of professional anti-drug community service，The investigator will adopt the Chinese traditional medicine JITAI combined with psychological intervention and social support for maintenance therapy after acute detoxification of the community of heroin addicts.The purpose is to observe the comprehensive treatment model to improve treatment compliance and relapse prevention，then the investigator will form a new model of community humane drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of The opioid dependence
* After detoxification.

Exclusion Criteria：

* Clinical Diagnosis of glaucoma and other severe mental disorder；
* serious organic disease within three months；
* can not comply with the test requirements；
* accept Hans therapy instrument；
* have tendence of suicide，self-injury and impulse；
* ECG abnormalities；
* ALT or AST greater than 5 times the upper limit of normal；
* history of epilepsy；
* Lactating or pregnant women，or women of childbearing age fails to take effective contraceptive measures；
* serious history of drug allergy or known allergy on traditional Chinese medicine JITAI；
* Study before the withdrawal less than a half-life of 5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The drug use pattern during observation period | Baseline ,26 weeks and 52 weeks
  The investigator will ues NHI(Nature History Interview) to describe the drug use pattern and and compare the different change among different groups during observation period

SECONDARY OUTCOMES:
The change of ASI(Addiction Severity Index) after the treatment and observation | Baseline,26weeks and 52 weeks
  The investigator will use ASI to describe the addiction severity of objects and compare the different change among different groups during observation period.
the change of drug use pattern during observation period | Baseline,26weeks and 52 weeks
  The investigator will ues NHI(Nature History Interview) to describe the drug use pattern and and compare the different change among different groups during observation period.
the change of SF-36(the MOS item short form health survey) after treatment and observation | Baseline,26 weeks and 52 weeks
  The investigator will use SF-36 to describe the health status of objects and compare the different change among different groups during observation period.
the change of SAS(Self-Rating Anxiety Scale) and SDS(Self-rating Depression Scale) during observation period | Baseline ,26weeks and 52 weeks
  The investigator will use SAS and SDS to describe the anxiety status and depression status then compare the different change among different groups during observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Min ZHAO, Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (2):
- China (2):
  - National Institute on Drug Dependence，Peking University, Beijing, Beijing Municipality
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan